CLINICAL TRIAL: NCT04132570
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of Intranasal Budesonide Aqueous Spray for Treatment of Rhinitis During Periods of High Airborne Pollution
Brief Title: A Study of Intranasal Budesonide Aqueous Spray for Treatment of Rhinitis During Periods of High Airborne Pollution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSURA001265; CCSURA001265 (Other: Johnson & Johnson Consumer, Inc., McNeil Consumer Healthcare Division); 5034003ALY4002 (Other: Johnson & Johnson Consumer, Inc., McNeil Consumer Healthcare Division)
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Rhinitis
Keywords: Airborne pollution; Rhinitis; Budesonide
MeSH Terms: conditions — Rhinitis | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide 256 mcg per Day (Treatment A) (Experimental): Participants will self-administer 2 nasal sprays of Budesonide (64 microgram [mcg]/spray) in each nostril once daily (every morning) up to 10 +\- 3 Days.
  Interventions: Drug: Budesonide
- Placebo (Treatment B) (Placebo Comparator): Participants will self-administer 2 nasal sprays of matching placebo in each nostril once daily (in the morning) up to 10 +\- 3 Days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Budesonide — Participants will self-administer 2 nasal sprays of Budesonide (64 mcg/spray) once daily up to 10 +\- 3 Days.
  Other Names: RHINOCORT
  Arms: Budesonide 256 mcg per Day (Treatment A)
Other: Placebo — Participants will self-administer 2 nasal sprays of matching placebo once daily up to 10 +\- 3 Days.
  Arms: Placebo (Treatment B)

SUMMARY:
The primary objective of this study is to assess the effectiveness of intranasal budesonide aqueous spray 256 microgram (mcg)/day for treatment of rhinitis symptoms during times of high airborne pollution.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported rhinitis symptoms triggered or worsened by airborne pollution, with agreement by physician at screening visit
* Participant must have moderate to severe rhinitis symptoms as defined by a 24-hour reflective total nasal symptom score (rTNSS) of at least 5 (maximum 9), based on three individual nasal symptom scores (nasal obstruction, secretion/runny nose, itching/sneezing) at the time of the screening visit, including at least one individual symptom score of 3 for nasal obstruction and/or secretion/runny nose
* Regularly have outdoor exposure during a normal week in the winter season, including greater than or equal to (>=) 1 hour on most days. Outdoor exposure may include commuting activities (such as walking/bicycle/auto/bus/city metro train travel), outdoor work, exercise, shopping, or other outdoor activities
* A woman of childbearing potential must have a negative urine pregnancy test (beta human chorionic gonadotropin [beta hCG]) at screening and agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after the last administration of study agent
* Male participants who are not surgically sterilized and are heterosexually active with a woman of childbearing potential, must agree to use a barrier method of contraception (example condom with spermicidal foam/gel/film/cream/suppository) and to not donate sperm during the study and for 30 days after last receiving study agent. Note that barrier methods must also be used in all male subjects sexually active with pregnant partners for at least 30 days after last study agent administration
* Participants can understand the questionnaires and are able to complete the questionnaires in the format provided
* Reside in the same city as the study site that they will be visiting

Exclusion Criteria:

* History of hypersensitivity to budesonide or any ingredients in the formulation
* Upper respiratory infection within 2 weeks of screening visit
* Current symptoms consistent with diagnosis of common cold, influenza, or other respiratory infection according to physician evaluation
* Using of N-95 masks days during with high airborne pollution
* Presence of nasal polyps or deviated septum as confirmed by nasal endoscopy
* History of nasal surgery
* Presence of chronic or active rhinosinusitis or sinusitis
* Systemic, intranasal or topical corticosteroid use within 1 month, intranasal or systemic decongestants within 3 days, antihistamine use within 1 week, intranasal cromolyn within 2 weeks, leukotriene use within 1 month, or immunotherapy within 2 years of screening visit
* Asthma, with the exception of mild intermittent asthma not requiring medication
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (example compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in 24-hour Reflective Total Nasal Symptom Score (rTNSS) | Baseline up to 10 days (24 hours each day)
  Mean change from baseline in 24-hour reflective total nasal symptom score (rTNSS) calculated as the sum of the participant-assessed 24-hour reflective severity ratings for three individual nasal symptom scores (nasal obstruction, secretion/runny nose, itching/sneezing) averaged over the first 10-day treatment period. Baseline value will be a single 24-hour rTNSS recorded on the no-treatment evening following the baseline visit. The individual nasal symptom scores will be recorded at home by participants in their diary on a four point scale (from 0=none to 3=severe). The sum of the individual scores will form the 24-hour rTNSS.

SECONDARY OUTCOMES:
Subject Global Impression of Change (SGIC) at the Final Efficacy Assessment | Day 10 (+/-3)
  Participant will rate Global Impression of Change at Final Efficacy Assessment on a 5-point scale from 0 (symptoms were aggravated) to 4 (total control over symptoms). An increase in score indicates the improvement in condition.
Mean Change from Baseline in Individual Nasal Symptoms Scores (NSS) | Baseline to 10 days (24 hours each day)
  Mean Change from Baseline in individual NSS for nasal obstruction, secretion/runny nose, and itching/sneezing averaged over the first 10-day treatment period will be reported using 4-point scale from 0=None, 1=Mild, 2=Moderate, or 3=Severe.
Mean Change from Baseline in 24-hour Reflective Individual non-Nasal Symptoms Score (Cough and Post-Nasal Drip) | Baseline to 10 days (24 hours each day)
  Mean Change from Baseline in 24-hour reflective Individual non-Nasal Symptoms Score for cough and post-nasal drip averaged over the first 10-day treatment period, using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe condition.
Number of Participants With Adverse Events (AEs) as a Measure of Safety | Up to Day 10 +/- 3 days or up to 30 days after the last day of the study treatment period (Day 10)
  An AE is any untoward medical occurrence in a clinical study subject administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — BEIJING TONGREN HOSPITAL, CMU; Chunguang Shan, Principal Investigator — THE SECOND HOSPITAL TO HEBEI MEDICAL UNIVERSITY; Weiwei Liu, Principal Investigator — Cangzhou Center Hospital; Guoji Zhang, Principal Investigator — BAODING FIRST CENTER HOSPITAL; Yaozhong Han, Principal Investigator — The No. 2 Hospital of Baoding; Yongjian Ma, Principal Investigator — THE NO.2 PEOPLE'S HOSPITAL OG WEIFANG; Guanggang Shi, Principal Investigator — Shandong Provincial Hospital
Locations (6):
- China (6):
  - Beijing Tongren Hospital, Cmu, Beijing, Beijing Municipality
  - The No.2 Hospital of Baoding, Baoding, Hebei
  - Cangzhou Center Hospital, Cangzhou, Hebei
  - The Second Hospital to Hebei Medical University, Shijiazhuang, Hebei
  - Shandong provincial hospital, Jinan, Shandong
  - The No.2 People'S Hospital Og Weifang, Weifang, Shandong

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSURA001265&attachmentIdentifier=71fdcdf6-82c9-48ba-960d-b9f6d9c3fe0a&fileName=CSR-Synopsis-5034003ALY4002-306308.pdf&versionIdentifier=